CLINICAL TRIAL: NCT04292483
Title: Pulmonary Capillary Recruitment With Pulmonary Vasodilator Therapy in Patients With Univentricular Heart Physiology and Failing Total Cavo-pulmonary Connection.
Brief Title: Pulmonary Capillary Recruitment in Fontan Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Tel Aviv University (Other); Old Dominion University (Other)
Responsible Party: Principal Investigator, Dr David Langleben, Professor of Medicine (Cardiology), Jewish General Hospital
Other Study IDs: 1900-5, 00-034
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Nitric Oxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nitric Oxide — Inhaled vasodilator to increase pulmonary capillary perfusion

SUMMARY:
This study evaluates the effects of pulmonary vasodilator therapy on pulmonary capillary blood flow by measuring the functional capillary surface area (FCSA) at baseline and post nitric oxide inhalation, through the injection of 3H-benzoyl-Phe-Ala-Pro (BPAP). FCSA will be related to flow and other hemodynamic parameters in order to determine if there is capillary recruitment or distention in Fontan patients. We will also compare baseline FCSA measurements with previously studied normal subjects, to assess the difference in hemodynamic pulmonary functional parameters between these single ventricle physiology patients and normal subjects.

ELIGIBILITY:
Inclusion Criteria:

Fontan failures will be defined as patients with single ventricle physiology and TCPC with clinical signs of dysfunction defined as any of the following:

1. Decreased functional class WHO/NYHA II or more and clinical signs of congestion (ascites, peripheral edema, increased JVP) and/or NT-proBNP > 399 pg/ml based on [17].
2. Age > 18 years
3. Known Fontan's increased pressures a. Fontan mean pressure of ≥15 mmHg and/or transpulmonary gradient ≥ 5 mmHg. b. Pulmonary vascular resistance ≥ 2 woods units. And/or supporting evidence of end-organ damage

1. Clinical or paraclinical evidence of liver congestion and/or fibrosis

a. Evidence in ultrasound or other imaging techniques of liver congestion and/or changes related to cardiac cirrhosis.

b. Fibroscan with grade 2 or + 2. Paraclinical signs of portal hypertension defined as 2 or more:

1. Thrombocytopenia defined as platelet count < 150.0000
2. Leukocytopenia defined as white blood cell less than 4.500
3. Esophageal varices on esophagoduodenoscopy.
4. Splenomegaly on imaging -

Exclusion Criteria:

1. Presence of fenestration - the shunts include veno-veno collaterals
2. Significant anemia defined as Hgb < 120 mg/dl
3. Pregnancy at the moment of the procedure.
4. Taking angiotensin-converting enzyme inhibitors or angiotensin receptor blockers.
5. Usage of nitrates, phosphodiesterase inhibitors or calcium blockers within 3 months of the study.

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with Fontan failure as described above
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional capillary surface area | 30 minutes
  Measurement of functional capillary surface area pre and post inhaled nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: David Langleben, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No